CLINICAL TRIAL: NCT03845946
Title: International Registry of Isolated Angioedema
Brief Title: CLOUD-R HAE REGISTRY
Acronym: CloudRHAE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.187
Record Dates: First submitted 2019-01-08; First posted 2019-02-19 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: ANGIOEDEMA
MeSH Terms: conditions — Angioedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Hereditary angioedema type I/II: Hereditary angioedema with C1Inh deficiency
  Interventions: Behavioral: angioedema
- Acquired angioedema: Angioedema with acquired C1Inh deficiency
  Interventions: Behavioral: angioedema
- Drug induced angioedema: Angioedema associated with ACEi used
  Interventions: Behavioral: angioedema
- Mast cell induced angioedema: Spontaneous mast cell induced isolated angioedema
  Interventions: Behavioral: angioedema
- Hereditary angioedema with nC1Inh: Hereditary angioedema with normal C1Inh and with F12, PLG, ANGPT2 mutations
  Interventions: Behavioral: angioedema

INTERVENTIONS:
Behavioral: angioedema — electronic tracking book

SUMMARY:
Angioedema is a disease characterized by the appearance of self-limiting edema that last 1-5 days and affect the subcutaneous tissue and/or gastrointestinal and oropharyngeal mucosa. In this last location edema can be lethal causing asphyxia, in all other cases full recovery is complete. Attacks can appear as part of the syndrome urticaria angioedema and can be of allergic origin. But there is a group of non-allergic angioedema that occur without hives and can be either hereditary or acquired. These angioedema are identified in some cases on the basis of etiology, in others are identified by the mediator and an overall classification of these forms of angioedema was published in 2014 as a result of a consent conference organized by the proponents of this registry. Being these forms of angioedema rare, there are not significative case studies inclusive of a high number of patients. This registry aims to collect in a single place a high number of subjects with recurring angioedema and without urticaria.

DETAILED DESCRIPTION:
The Grenoble center is the registry coordinator at the national level. It will contract directly with the Cloud R Company and will be in charge of coordinating the associated centers. It will therefore send the necessary documents for the good execution of the study, will ask each center to respect the current French regulatory, will organize and finance the set-up of the register in the associated centers.

The coordinating center will also centralize requests for data, publications or creation of additional eCRF pages of associated centers. It will be able to organize a national scientific committee every 6 months. It will thus be the link between the French centers, the scientific committee of the registry and the company Cloud R.

The coordinating center will also be responsible for enter and reliability of patient data from it center, as well as the associated centers.

Role of associated centers Associated Centers will be responsible for capturing and data reliability of their patients in eCRF, they will also create a personal account for each patient so that it can download the application "cloud R HAE carnet de suivi".

Investigators referent patient will have validated at each visit or after contact with the patient crisis returned to the patient via it electronic diary.

Associated Centers will keep informed twice a year the coordinator center of the state of inclusions in the register.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with isolated angioedema without associated wheals.
* Patients with hereditary angioedema with or without C1 deficiency.
* Major patient with consent (signature)
* Minor patient whose parents / legal guardians have given their consent (signature)

Exclusion Criteria:

* Patient unable to give consent.
* Wheals with angioedema

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with isolated angioedema without associated wheals
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Demographic patient data | 5 years
  Sexe and age of patient
Clinical characteristics | 5 years
  summary of patient visit report
Comorbidity | 5 years
  additional diseases
Angioedema diagnosis | 5 years
  type of angiodema
Angioedema diagnosis | 5 years
  position of genetic mutation if applicable
Angioedema diagnosis | 5 years
  biology marker : C1inh, C4, C1q, anti C1inh
Angioedema diagnosis | 5 years
  family history
Duration and severity of acute angioedema events | 5 years
  start date
Duration and severity of acute angioedema events | 5 years
  localization
Duration and severity of acute angioedema events | 5 years
  time before treatment
Duration and severity of acute angioedema events | 5 years
  time to resolution
Duration and severity of acute angioedema events | 5 years
  need access to hospital
Treatments used in managing the acute angioedema event | 5 years
  name
Treatments used in managing the acute angioedema event | 5 years
  dose
Treatments used in managing the acute angioedema event | 5 years
  date and time of acute treatment
Treatments used in the prophylaxis of angioedema | 5 years
  name
Treatments used in the prophylaxis of angioedema | 5 years
  dose
Treatments used in the prophylaxis of angioedema | 5 years
  start date

CONTACTS AND LOCATIONS:
Overall Officials: laurence bouillet, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, Isere, France

IPD SHARING:
Plan to Share IPD: No